CLINICAL TRIAL: NCT05981794
Title: The Effects of a Heating Pad on Anxiety, Pain, and Distress During In-office Cystoscopy and Urodynamics: a Randomized Controlled Trial
Brief Title: Heating Pad for in Office Cystoscopy and Urodynamic Testing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution and changed to new PI, there was no funding secured for this study.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC20230455H
Record Dates: First submitted 2023-07-22; First posted 2023-08-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Pain; Distress, Emotional
Keywords: Cystoscopy; Urodynamic study
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 manner to the treatment group (those receiving a heating pad with heat during the procedure) or control group (those who receive a heating pad without heat). The study is prospective, and randomization will be performed by a random allocation table. Randomization will be stratified by sex, procedure, and provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Heating Pad heated (Experimental): An electrical heating pad will be applied prior to the cystoscopy or urodynamic procedure
  Interventions: Device: Electrical heating pad
- Placebo heating pad (Placebo Comparator): An electrical heating pad that is not heated will be applied prior to the cystoscopy or urodynamic procedure
  Interventions: Device: Sham heating pad

INTERVENTIONS:
Device: Electrical heating pad — A powered heating pad
  Other Names: Heating pad
  Arms: Heating Pad heated
Device: Sham heating pad — A heating pad that is not powered on
  Other Names: Non-heated heating pad
  Arms: Placebo heating pad

SUMMARY:
Patient frequently report experiencing discomfort associated with cystoscopy or urodynamic studies (UDS), and a small percentage of patients refuse these important procedures due to discomfort or fear of discomfort. Heating pads are an inexpensive and low-risk way to reduce patient discomfort during these procedures, which to our knowledge has not been investigated in the United States.

DETAILED DESCRIPTION:
Invasive office procedures such as cystoscopy and urodynamic studies (UDS) are commonly performed for many urologic and Urogynecologic conditions including, but not limited to, incontinence, voiding dysfunction, urinary retention, hematuria, and other lower urinary tract symptoms. Cystoscopy involves the insertion of a rigid or flexible cystoscope through the urethra and into the bladder. Urodynamic studies involve the placement of urethral and rectal catheters. Both cystoscopy and UDS involve filling the bladder with fluid, and these procedures are essential to the diagnosis and management of many of the conditions listed above.

While both procedures are office procedures that are generally well tolerated, some patients can experience significant discomfort, pain, or anxiety. Some nonpharmacologic therapies have been investigated to relieve anxiety, pain, and distress, such as music and aromatherapy. Heating treatments are also known to reduce muscle pain by increasing local blood flow and decreasing distress. The use of a heating pad has become an established complementary modality in some invasive procedures. A previous study from South Korea has shown benefit of heating pad use for anxiety, pain, and distress during cystoscopy and UDS; however to our knowledge, there are no studies evaluating the effect of heating pad use on patients in the United States, who may have inherent demographical differences compared to patients from South Korea.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to give informed consent
* Able to read and write English or Spanish

Exclusion Criteria:

* Refusal to participate
* Contraindications to cystoscopy or urodynamic testing
* Patients who receive other procedures or treatment at the time of cystoscopy, such as bladder biopsy or Botox injection
* Patients with spinal cord injury or lack of sensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety visual analog scale (VAS) | Pre- and Post-procedure (about 30 minutes)
  Change in score on a 10-point visual analog scale where where 0 indicates the least amount of anxiety and 10 the greatest
Hospital Anxiety and Depression Survey (HADS) | Pre- and Post-procedure (about 30 minutes)
  Change in score on the anxiety subscale score, a total score of 0-21 is possible, with a score between 0-7= Normal, 8-10= Borderline abnormal and 11-21= abnormal
Change in Pain (VAS) | Pre- and Post-procedure (about 30 minutes)
  Change in score on a visual analog scale (VAS) from 0-10, where 0 indicates the least amount of pain and 10 the greatest
Change in Distress (VAS) | Pre- and Post-procedure (about 30 minutes)
  Change in score on a visual analog scale (VAS) from 0-10, where 0 indicates the least amount of distress and 10 the greatest
Blood pressure measure | Pre- and Post-procedure (about 30 minutes)
  Change in blood pressure
Heart rate | Pre- and Post-procedure (about 30 minutes)
  Change in heart rate

SECONDARY OUTCOMES:
Wait time | Pre-procedure to beginning of procedure (about 30 minutes)
  Amount of time spent waiting prior to procedure
Time spent on procedure | Pre- to Post-procedure (about 30 minutes)
  Amount of time taken to complete procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Tibon, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: When summary data are published or otherwise made available at study completion